CLINICAL TRIAL: NCT06369363
Title: Estrogen Deficiency on Cardiovascular Risk: Sympathetic Responses and Pro-inflammatory Cytokines
Brief Title: Estrogen Deficiency on Cardiovascular Risk
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Milton S. Hershey Medical Center (Other)
Responsible Party: Principal Investigator, Lu Qin, Assistant Professor in Department of Medicine, Milton S. Hershey Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: STUDY000024245
Record Dates: First submitted 2024-04-11; First posted 2024-04-17 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Postmenopausal Symptoms; Cardiovascular Diseases
MeSH Terms: conditions — Cardiovascular Diseases | interventions — Estradiol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Estradiol (Experimental)
  Interventions: Drug: Estradiol

INTERVENTIONS:
Drug: Placebo — Subjects will be assigned to 1 week of transdermal placebo patch.
  Arms: Placebo
Drug: Estradiol — Subjects will be assigned to 1 week of transdermal estradiol (0.05 mg/day) patch.
  Arms: Estradiol

SUMMARY:
To explore how estrogen deficiency impacts the blood pressure (BP) and sympathetic nerve activity (SNA), and how it impacts the production of the key pro-inflammatory mediators such as Tumor necrosis factor α (TNF-α), interleukin-1β (IL-1β), and interleukin-6 (IL-6). It is hypothesized that estrogen deficiency increases BP, SNA and the pathway activities of the key pro-inflammatory mediators. Those effects are impacted through the downregulation of the estrogen receptor.

DETAILED DESCRIPTION:
In the United States, cardiovascular disease (CVD) is one of the major health concerns and affects approximately 6.5 million people over 40. As the number of elderly women increases, CVD becomes an increasing problem. Estrogen is cardioprotective, and the menopause condition in the aging female population induces the loss of this protective effect. There has been a dilemma for medical treatment in CVD patients with comorbidities including endometriosis or breast cancer history. Overall, these patients lose the cardioprotective effect of estrogen and increase the risk of CVD development. However, there is still little understanding regarding the mechanism for how estrogen suppression in women accelerates CVD development. The proposed studies are, therefore, the essential first step to elucidating how estrogen alters mechanisms underlying CVD and provide the preclinical data to design studies for future alternative intervention strategies for CVD patients undergoing estrogen suppression therapies.

ELIGIBILITY:
Inclusion Criteria:

* Age 54-75 years
* Healthy participants who are capable of giving informed consent
* Classified as postmenopausal or stop having period >1year or had a full hysterectomy surgery
* Any race or ethnicity
* Have satisfactory history and physical exam
* Free of acute medical conditions

Exclusion Criteria:

* <54 or >75 years
* Medications that could alter cardiovascular, thermoregulatory, or peripheral vascular control (e.g. Angiotensin converting enzyme inhibitors, statins, beta blockers, etc.);
* Self-reported history of long-term menstrual irregularities, vaginal bleeding, or other gynecological conditions that could influence study outcomes
* Use of hormone therapy during 6 months prior to study enrollment
* Allergy to latex
* Current smoker
* Have any clinically relevant history or the presence of metabolic (e.g., diabetes), respiratory, renal, hepatic, gastrointestinal, hematological, lymphatic, neurological, cardiovascular, or other disease or diseases that, in the opinion of the research team, exclude the subject from participation.
* Presenting with a resting blood pressure of 150/100 or higher
* Contraindications to a maximal exercise test or an indication for early termination of an exercise test
* Taking any medications that affect vascular control or autonomic function (e.g. beta blockers, ACE inhibitors, calcium channel blockers, etc.)
* Contraindications to estrogen patch: include undiagnosed vaginal bleeding; known, suspected, or history of breast cancer; known or suspected E2-sensitive neoplasm; history of deep venous thrombosis or pulmonary embolism; current or recent arterial thromboembolic disease; liver dysfunction and disease; known or suspected pregnancy.
* Past/current history of venous thromboembolism, hypercoagulation or thrombopenia
* Past/current history of hormone-responsive cancer
* Past/current history of endometrial hyperplasia
* Patient has a recent drug or alcohol abuse history (less than 6 months) or is currently using or abusing excessive alcohol or drugs. Excessive alcohol will be defined as greater than 14 drinks per week.

Ages: 54 Years to 75 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-09 (Estimated); Primary Completion 2028-09 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Red blood cell flux | Recorded continuously for up to 4 hours during the study visit
  Percentage relative to the maximum flux level
Mean arterial pressure (mmHg) | Recorded continuously for up to 4 hours during the study visit
  Calculated from the systolic and diastolic blood pressure
baseline plasma TNF-α concentration (pg/ml) | Upon participants' arrival to the first study visit up to 5 minutes
  Measured by ELISA kits
One week post-intervention plasma TNF-α concentration (pg/ml) | Upon participants' arrival to the second study visit (1 week after the first visit)
  Measured by ELISA kits
baseline plasma IL-1β concentration (pg/ml) | Upon participants' arrival to the first study visits up to 5 minutes
  Measured by ELISA kits
One week post-intervention plasma IL-1β concentration (pg/ml) | Upon participants' arrival to the second study visit (1 week after the first visit)
  Measured by ELISA kits
baseline plasma IL-6 concentration (pg/ml) | Upon participants' arrival to the first study visits up to 5 minutes
  Measured by ELISA kits
One week post-intervention plasma IL-6 concentration (pg/ml) | Upon participants' arrival to the second study visit (1 week after the first visit)
  Measured by ELISA kits

SECONDARY OUTCOMES:
baseline plasma estrogen (pg/ml) | Upon participants' arrival to the first study visits up to 5 minutes
  Measured by ELISA kits
One week post-intervention plasma estrogen (pg/ml) | Upon participants' arrival to the second study visit (1 week after the first visit)
  Measured by ELISA kits

CONTACTS AND LOCATIONS:
Overall Officials: Lu Qin, PhD, Principal Investigator — Penn State College of Medicine